## **Patient Informed Consent Form for Study Participation**

| Study Title: | Genetic Determinants of the Coronary Microvascular |
|---|---|
| | Obstruction in Percutaneous Coronary Interventions |
| Protocol Number: | CMVO-SNP-2022 |
| Study Number: | NCT05355532 |
| Document date and | Version number 1 from April 24, 2022 |
| version: | |
| Sponsor: | Privolzhsky Research Medical University |
| Principal | Principal Investigator: |
| Investigator: | Ilya Grigorievich Pochinka, MD |
| | Research Center: |
| | State Budgetary Healthcare Institution of Nizhny Novgorod |
| | Region "City Clinical Hospital No. 13 of Avtozavodsky |
| | District of Nizhny Novgorod" |
| | Research Center Address: |
| | 51 Patriotov Street, Avtozavodsky District, |
| | Nizhny Novgorod, Russian Federation, 603018 |
| | Research Center Phone: |
| | +7 (831) 255-28-80 |

You are being offered the opportunity to participate in this genetic study because you have been diagnosed with myocardial infarction and have undergone percutaneous coronary intervention. During this procedure, you \_\_\_\_ developed coronary microvascular obstruction. Below is a brief description of the study and your role as a potential participant. Please read this information carefully and ask the investigator any questions you may have to make an informed decision about participating in the study.

You are not obligated to participate in this study. Your decision will not affect your future treatment. Regardless of your choice, you will receive all necessary medical care in full. Participation in the study is free of charge.

The purpose of the study is to investigate genes associated with the development of coronary microvascular obstruction during percutaneous coronary interventions. If you agree to participate, a blood sample will be taken from you for genetic testing.

This study does not involve any special therapy or medical interventions other than the blood draw for genetic analysis. The blood sample (2 mL) will be collected once from a peripheral vein in the operating room where you are currently located after the percutaneous coronary intervention. Before the blood draw, you must sign this informed consent form.

Since the study does not involve medication or medical procedures (except for a standard venous blood draw), it carries no clinical risks and is not associated with the risk of side effects or adverse reactions.

Participation in the study will provide valuable medical information about the course of myocardial infarction and help your doctor determine the optimal treatment strategy to improve your prognosis.

This study can only be conducted by collecting and using your medical information. Data protection laws grant you the right to control the use of your personal information. By signing this form, you grant special permission for the verification, transfer, and processing of your information as follows:

- Doctors conducting the study, the ethics committee, and regulatory inspectors may review your medical information through direct access.
- Research data may be used and shared for legally permitted research and scientific purposes.

The study has been approved by the local ethics committee.

| Patient study number | | - | |
|----------------------|------------|---|-----------------|
| Patient | | | |
| Date: "" | 20 Time: " | : | _" Signature: _ |
| Physician | | | |
| Date: "" | 20 Time: " | : | _" Signature: |